CLINICAL TRIAL: NCT05513560
Title: REcovering From COVID-19 Lingering Symptoms Adaptive Integrative Medicine (RECLAIM)
Brief Title: RECLAIM: Recovering From COVID-19 Lingering Symptoms Adaptive Integrative Medicine
Acronym: RECLAIM
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: We are analyzing data for efficacy
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21-6203
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-02

CONDITIONS: Long COVID; Post COVID Condition; Post Acute Sequelae of COVID-19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — ibudilast; Pentoxifylline

STUDY DESIGN:
Intervention Model Description: RECLAIM is a Canada-wide phase ll/lll, prospective, adaptive randomized controlled platform trial that is intended to study various interventions for patients with long COVID. Interventional arms may be discontinued based on interim analysis results and new interventions may be selected and included as part of the platform as the trial progresses. As such, the protocol and consent documents are a modular design including;
  * Master Protocol and informed consent documents: Contain information applicable to the whole platform.
  * Interventional Sub-Protocols: Contain additional information, specific to the interventional arm.
  Interventional Sub-Protocols may be modified, discontinued, or added without revisions to the Master Protocol.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants are blinded to intervention in so far as the labelling of the study intervention. However, it is possible that the participant may figure out allocation arm, by the mode of administration, dosing frequency (once a day versus 3 times per day), and treatment form (pill, powder, intervention) etc.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- IBUDILAST (Experimental): Participants will receive 20 mg dose (2 pills) twice per day taken by mouth.
  Interventions: Drug: Ibudilast
- PENTOXIFYLLINE (Experimental): Participants will receive a 400mg dose (1 pill) 3 times per day taken by mouth.
  Interventions: Drug: Pentoxifylline
- PLACEBO (Placebo Comparator): Participants will receive 2 placebo pills twice per day taken by mouth OR 1 placebo pill 3 times a day taken by mouth.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ibudilast — 10mg pills, 2 pills twice per day
  Other Names: MN-166
  Arms: IBUDILAST
Drug: Pentoxifylline — 400mg pill 3 times per day
  Arms: PENTOXIFYLLINE
Other: Placebo — Placebo matching ibudilast, 2 pills twice per day OR placebo matching pentoxifylline 1 pill 3 time per day.
  Arms: PLACEBO

SUMMARY:
The researchers propose to develop a Canada-wide, adaptive randomized clinical platform trial to assess the effectiveness of various interventions in patients with lingering symptoms of COVID-19 ("Long COVID"). Participants will be randomized initially to 1 of 3 arms, including placebo (control) and 2 interventions. Because this is an adaptive trial, arms can be dropped if found to be ineffective and new arms can be added.

Interventions will last for 2 months and participants will be followed for an additional 4 months (6 months total). Approximately 800-1000 patients with Long COVID will be recruited across Canada. Results from this trial will accelerate the availability of high-quality, real-time evidence and solutions to enable Canada to improve the clinical care of patients with Long COVID.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Positive COVID-19 test by nasopharyngeal swab RT-PCR (reverse transcription polymerase chain reaction) test, antibody or antigen tests at least 3 months prior to randomization; OR Presumed COVID-19 assessed by the site investigator (no positive COVID-19 test) with acute illness after October 15, 2019.
3. Patients should be treated with standard of care therapies (as discussed in the study manual) for at least 4 weeks prior to entry into trial.
4. Lingering COVID-19 symptoms beyond 3 months from onset of acute COVID and symptoms have lasted at least 2 months. The onset of COVID is considered the earliest of two dates: the date of positive test or the date of first symptoms;
5. Lingering symptoms from COVID-19 present at the time of randomization.
6. Female patients of childbearing potential (as assessed by the overseeing Investigator) who are sexually active must agree to practice true abstinence or use effective methods of contraception while on study treatment. Effective methods of contraception must be discussed and approved by the overseeing Investigator.
7. Must be able to provide informed consent and both willing and able to comply with study requirements.

Exclusion Criteria:

1. Patients who had mechanical ventilation or extracorporeal membrane oxygen (ECMO) for COVID-19;
2. Current end-organ failure, organ transplantation, or current hospitalization in acute care hospital;
3. Contraindications to all of the study interventions;
4. Co-enrolment in another interventional trial (co-enrolment in an observational study is permitted);
5. Currently pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
SF-36 physical component score (PCS) | from baseline to two months
  mean change in the SF-36 (v.1) physical component score (PCS)

SECONDARY OUTCOMES:
Symptoms scale | Baseline/Randomization weekly to 2 months, then once monthly to 6 months.
  Three point Likert scale assessing how bothersome symptoms are on a weekly basis for two months then monthly until end of study, as reported by the participant: to provide a granular, detailed picture of the symptom trajectory.
Symptom Checklist | Baseline/Randomization weekly to 2 months, then once monthly to 6 months.
  Symptom Checklist (adapted from the De Paul Symptom Questionnaire (DSQ2), the World Health Organization Global COVID-19 Clinical Platform's Post COVID-19 CRF and the Symptom Burden Questionnaire for Long COVID): to track symptom trajectory.
Six Minute Walking Test (6MWT) with oximetry | Baseline/Randomization and 2 months
  Subjects walk as far as they can in six minutes while receiving maximum encouragement. It is simple to execute, inexpensive, standardized and gives a tangible measure of functional exercise capacity. It has been validated in many different populations. The 6MWT will be conducted according to American Thoracic Society standards.
TestMyBrain cognitive testing | Baseline/Randomization to 1, 2 months 3 and 6 months
  TestMyBrain was developed as a tool to collect large, population-based samples for understanding the relationship between cognition, emotion, social functioning, and health. This test battery will take about 20 minutes to complete and will assess: verbal, episodic and working memory, attention, processing speed, basic psychomotor response speed, and cognitive control.
Post COVID19 functional status scale | Baseline/Randomization to 1, 2 months 3 and 6 months
  The post-COVID-19 functional status (PCFS) scale focuses on relevant aspects of daily life during follow-up after the infection. The scale is intended to help users become aware of current functional limitations in COVID-19 patients, whether or not as a result of the specific infection, and to objectively determine this degree of disability. The scale is ordinal, has 6 steps ranging from 0 (no symptoms) to 5 (death), and covers the entire range of functional outcomes by focusing on limitations in usual duties/activities either at home or at work/study, as well as changes in lifestyle. The PCFS demonstrates good construct validity.
Reintegration to Normal Living Index (RNLI) | Baseline/Randomization to 1, 2 months 3 and 6 months
  This short self-administered assessment tool will determine the degree to which participants reintegrate into normal social activities such as recreation, mobility in the community and interaction in family and other relationships. This tool has been validated in community living adults with mobility limitations.
Fatigue Scale | Baseline/Randomization to 1, 2 months 3 and 6 months
  The Fatigue Scale was adapted from the De Paul Symptom Questionnaire (DSQ2)'s 38 questions assessing medical history of Myalgic Encephalitis/Chronic Fatigue Syndrome (ME/CFS), comorbidities, medications, impact on quality of life and daily activities, etc.
Brief Fatigue inventory | Baseline/Randomization to 1, 2 months 3 and 6 months
  The self-administered Brief Fatigue Inventory is composed of 9 items evaluated on a 10-point scale, assessing severity of fatigue and impact of fatigue on daily life. It takes approximately 2-3 minutes to complete.
Post-Exertional Malaise | Baseline/Randomization to 1, 2 months 3 and 6 months
  The self-administered DPEMQ is comprised of three sections assessing post-exertional malaise (PEM): (i) onset and triggers of PEM (9 questions), (ii) consequences and symptoms (14 questions), (iii) duration, recovery and pacing (7 questions).
Mental Health - Post-traumatic Stress Disorder Checklist (PCL-5) | Baseline/Randomization to 1, 2 months 3 and 6 months
  The PCL-5 is a validated, reliable, 20-item self-report measure that assesses the 20 Diagnostic and Statistical Manual 5 (DSM-5) symptoms of Post-Traumatic Stress Disorder (PTSD). It takes approximately 5-10 minutes to complete.
Mental Health - General Anxiety Assessment Form (GAD-7) | Baseline/Randomization to 1, 2 months 3 and 6 months
  The GAD-7 is a valid and efficient tool for screening for generalized anxiety disorder and assessing its severity in clinical practice and research. It is an easy-to-use, self-administered patient questionnaire that can be completed in minutes.
Mental Health - Patient Health Questionnaire (PHQ-9) | Baseline/Randomization to 1, 2 months 3 and 6 months
  The PHQ-9 is a validated, multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression. It incorporates Diagnostic and Statistical Manual 1V (DSM-IV) depression diagnostic criteria with other leading major depressive symptoms into a brief self-report tool. The PHQ-9 is brief and useful in clinical practice.
  The PHQ-9 is completed by the patient in minutes and is rapidly scored by the clinician. The PHQ-9 can also be administered repeatedly, which can reflect improvement or worsening of depression in response to treatment.
Mental Health Composite score (MCS) of the SF-36 | Baseline/Randomization to 1, 2 months 3 and 6 months
  The self-administered SF-36 evaluates eight health concepts: physical functioning, role functioning-physical, bodily pain, general health, vitality, social functioning, role functioning-emotional, and mental health. Previous studies have used this instrument in many different populations and it takes approximately 15 minutes to complete.
Dyspnea | Baseline/Randomization to 1, 2 months 3 and 6 months
  Assessed using the Borg Dyspnea scale. This short assessment tool assesses perceived shortness of breath on exertion using a 10 point scale as assessed by the patient.
Blood samples | Baseline/Randomization and 2 months
  Blood samples will be used in correlative studies using advanced multi-omic and machine learning methods to better understand our results so as to identify phenotypes that will benefit from specific therapies

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Cheung, MD,PhD, Principal Investigator — University Health Network, Toronto; George Tomlinson, PhD, Principal Investigator — University Health Network, Toronto; Peter Juni, MD, PhD, Principal Investigator — Oxford University, UK
Locations (3):
- Canada (3):
  - The Ottawa Hospital, Ottawa, Ontario
  - University Health Network, Osteoporosis Department, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No